CLINICAL TRIAL: NCT05362344
Title: A Multi-Center Study of Non-Invasive Colorectal Cancer Evaluation in Cystic Fibrosis (NICE-CF)
Brief Title: Colorectal Cancer Screening in Cystic Fibrosis
Acronym: NICE-CF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington, the Collaborative Health Studies Coordinating Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NICE-CF
Record Dates: First submitted 2022-04-28; First posted 2022-05-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis; Colorectal Cancer; Adenoma
Keywords: Cystic Fibrosis; Colorectal Cancer; Cancer screening; Adenoma
MeSH Terms: conditions — Cystic Fibrosis; Colorectal Neoplasms; Adenoma | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NICE-CF Cohort: Adults with CF ages 18 - 75 years who are due for a routine screening or surveillance colonoscopy for colon cancer.
  Interventions: Procedure: Stool tests

INTERVENTIONS:
Procedure: Stool tests — Non-invasive, stool-based tests for colorectal cancer screening.
  Other Names: Stool-based Fecal Immunochemical Testing (FIT) test and Stool-based DNA test (Cologuard) test.

SUMMARY:
This multi-center study will compare multi-target DNA and quantitative FIT stool-based testing to colonoscopy in individuals with Cystic Fibrosis (CF) undergoing colon cancer screening with colonoscopy. The primary endpoint is detection of any adenomas, including advanced adenomas and colorectal cancer (CRC).

DETAILED DESCRIPTION:
NICE-CF is a cross-sectional, multi-center study comparing stool-based testing (multi-target DNA test and quantitative FIT test) to standard of care colonoscopy for colorectal cancer (CRC) screening in people with CF. The study includes an enrollment visit, two stool samples completed at home, a clinical screening colonoscopy, and three participant surveys which will be completed at enrollment or remotely.

The total duration of participant participation will be 3-12 months, depending on the timing of the completion of the stool samples and the participant's colonoscopy. The targeted participant timeline is 3 months from enrollment to the completion of a clinical screening colonoscopy. To allow for varying site-specific clinical colonoscopy scheduling delays and COVID delays in scheduling, the duration of time between submitting stool samples and screening colonoscopy may extend up to 12 months for inclusion of data in the study. However, participating sites must notify the DCC to obtain preapproval for greater than 3 months duration between stool-based testing and colonoscopy.

CF patients who are eligible for CRC screening will either be enrolled during an in-person CF clinic visit or via phone/video if clinic visits are taking place remotely. Participants will be asked to perform stool sample collection at home, and then complete their colonoscopy within three to twelve months of submission of the stool sample.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with CF ages 18 - 75 years and due for a routine screening or surveillance colonoscopy for colon cancer
2. Cystic Fibrosis diagnosis, defined by a sweat chloride test result ≥ 60 mmol/L (may be of historic value), and/or documented CF-causing CFTR mutations and clinical features of CF
3. Capable of understanding the purposes and risks of the study in English or Spanish and willing to participate and sign informed consent
4. Referred for screening or surveillance colonoscopy for CRC (current standard of care) and willing to undergo colonoscopy and stool testing
5. Able to access the Internet to complete self-administered surveys

Exclusion Criteria:

1. Any condition that, in the opinion of the site PI, introduces undue risk by participating in this study
2. Incapable of understanding the purposes of the study or informed consent for any reason
3. Pregnancy
4. Active inflammatory bowel disease as defined by a prior diagnosis of Crohn's Disease or Ulcerative Colitis, based on both clinical and histopathologic findings and the individual currently on medical therapy for Crohn's disease or Ulcerative Colitis.
5. Personal history of colon cancer diagnosis and treatment within 5 years of enrollment
6. Symptoms that merit colonoscopy for diagnostic purposes rather than as screening for CRC
7. Known history of familial colon cancer syndrome that has been confirmed by previous genetic testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18-75 with cystic fibrosis (CF) eligible for routine colon cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of multi-target stool DNA test and quantitative fecal immunochemical (FIT) test | 3-12 months
  Negative predictive value (NPV) and sensitivity for detection of any adenomas, advanced adenomas, and CRC in stool-based testing.

SECONDARY OUTCOMES:
Specificity of multi-target stool DNA test and quantitative fecal immunochemical (FIT) test | 3-12 months
  Specificity and positive predictive value (PPV) of stool-based testing for any adenomas, advanced adenomas, and CRC

OTHER OUTCOMES:
Adenomas | 3-12 months
  Overall prevalence of any adenomas detected by screening and by colonoscopy
Advanced adenomas | 3-12 months
  Overall prevalence of advanced adenomas detected by screening and by colonoscopy
CRC detection | 3-12 months
  Overall prevalence of CRC detected by screening and by colonoscopy
Sessile serrated lesions | 3-12 months
  Overall prevalence of sessile serrated lesions detected by screening and by colonoscopy
Stool-based test feasibility | 3-12 months
  Proportion of patients who complete stool-based testing
Colonoscopy feasibility | 3-12 months
  Proportion of study participants who complete colonoscopy and stool-based testing
Comparison of multi-target stool DNA test and quantitative fecal immunochemical (FIT) test to detect any adenomas, advanced adenomas, and CRC in PwCF | 3-12 months
  Comparison of the predictive ability of the two tests
Ease of stool testing | 3-12 months
  Qualitative surveys on ease of stool sample collection and colonoscopy prep

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hachem, MD, Principal Investigator — St. Louis University; Sarah Jane Schwarzenberg, MD, Principal Investigator — University of Minnesota; Steven D. Freedman, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (26):
- United States (26):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - National Jewish Health, University of Colorado, Denver, Colorado
  - University of Miami Hospital, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - North Carolina Children's Hospital / UNC, Chapel Hill, North Carolina
  - Atrium Health Pulmonary Care, Charlotte, North Carolina
  - University Hospitals Rainbow Babies & Children's, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No